CLINICAL TRIAL: NCT02902445
Title: Glycan Attachment Specificity, Toward ROtavirus Vaccine IMprovement GASTROVIMc (Clinical Investigation) Evaluation of Individual Genetic Susceptibility in Severe Gastro-enteritis Rotavirus: Role of HBGA Polymorphisms & Biotechnology Improvement of RVA Vaccines
Brief Title: Glycan Attachment Specificity, Toward ROtavirus Vaccine IMprovement GASTROVIMc (Clinical Investigation)
Acronym: Gastrovimc
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0329
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2021-04

CONDITIONS: Gastroenteritis; Acute Gastroenteritis
Keywords: Vaccine; Polymorphism
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case group: 250 children from Nantes University Hospital and 150 children from Guyana Hospital admitted in paediatric emergency unit for diagnosed rotavirus acute gastroenteritis: rotavirus rapid screen test and oral swab for polymorphism exploration
  Interventions: Biological: rotavirus rapid screen test; Genetic: polymorphism exploration
- Control group: 250 children from Nantes University Hospital and 150 children from Guyana Hospital admitted in paediatric emergency unit without signs of infection and / or digestive clinical picture evocative of gastroenteritis.
  Paired with a case upon ethnicity or origin if impossible to match the ethnicity of the case.
  oral swab for polymorphism exploration
  Interventions: Genetic: polymorphism exploration

INTERVENTIONS:
Biological: rotavirus rapid screen test — According to routine care
  Groups: Case group
Genetic: polymorphism exploration — from an oral swab collected after parents consent

SUMMARY:
The GASTROVIM research explores the links between individual genetic susceptibility, genetic variability of rotavirus strains and effectiveness of immunization with the rotavirus vaccination: a clinical investigation to assess glycan attachment specificity, toward rotavirus vaccine improvement.

DETAILED DESCRIPTION:
The work will be carried out in France and in a tropical area of population with diverse geographical origins: the Guyana populated with Native Americans, people of European descent, people of Asian (Hmong) and a large source population African.

The first aim of the project will be to characterize the specificity of the VP8 * HBGA of RotaTeq and Rotarix vaccines in order to ensure their binding characteristics glycans are similar to those of recent P8 clinical strains circulating in France and were maintained in the culture passages.

The second objective will be to validate the impact of recently described polymorphisms HBGAs on susceptibility to infection by RVA through GASTROVIMc prospective clinical research.

The third objective will be to determine the relative role of recognition and HBGAs ganglioside in the initial attachment and viral entry.

The expression of HBGAs and ganglioside by permissive cell lines in culture human stem RVA be manipulated to define the role of glycans in attachment and infection.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 16.
* giving consent to participate if applicable (>6yo)
* Parents informed and written consent obtained
* admitted in paediatric emergency for wether an acute gastroenteritis (case group) or anything else than an infection or gastroenteritis (control group)

Exclusion Criteria:

* case group: rotavirus rapid screen test negative; viral gastroenteritis other than rotavirus; bacterial gastroenteritis
* control group: Family and / or patient unable to full informed consent to research; Infectious Pathology context in general.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 400 children admitted to the pediatric emergency for acute gastroenteritis (cases) and 400 children admitted to the pediatric emergency without evocative picture of infection or gastroentieritis
Sampling Method: Non-Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Absence / Presence of non-secretory polymorphisms FUT2- and Lewis Negative FUT3- | 6 months after inclusion

SECONDARY OUTCOMES:
Population frequency of new protective genotypes to rotavirus infection | Six months after inclusion
Absence / presence of genetic polymorphisms --other (Including FUT2- and FUT3-) | Six months after inclusion
Absence / presence of different viral strains Rotavirus (RVA) involved in the acute gastroenteritis episodes in French Guiana | Six months after inclusion
Absence / presence of various HBGA polymorphisms involved in acute gastroenteritis episodes in French Guiana | Six months after inclusion
population frequency of different etiologies of acute gastroenteritis viral, bacterial and / or parasitic (Cayenne) | Six months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christèle GRAS-LEGUEN, MD PhD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided